CLINICAL TRIAL: NCT06581328
Title: A Phase 4 Study Evaluating Moderate to Severely Active Ulcerative Colitis or Crohn's Disease and the Use of Vedolizumab Subcutaneous Within a Community Setting
Brief Title: A Study of Vedolizumab in Adults With Ulcerative Colitis or Crohn's Disease in the Community Setting
Acronym: PANORAMA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-4063
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- UC Participants: Vedolizumab (Experimental): Participants with moderate to severely active UC will receive vedolizumab 300 milligrams (mg), intravenous (IV) infusion at Weeks 0 and 2. Following the first 2 vedolizumab IV doses, participant may be switched to vedolizumab 108 mg subcutaneous (SC) injection at Week 6, to be administered every 2 weeks until Week 50. Treating health care practitioner (HCP) may give an additional dose of vedolizumab IV at Week 6 with mandatory transition by Week 14.
  Interventions: Drug: Vedolizumab IV; Drug: Vedolizumab SC
- CD Participants: Vedolizumab (Experimental): Participants with moderate to severely active CD will receive vedolizumab 300 mg, IV infusion at Weeks 0 and 2. Following the first 2 vedolizumab IV doses, participant may be switched to vedolizumab 108 mg SC injection at Week 6, to be administered every 2 weeks until Week 50. Treating HCP may give an additional dose of vedolizumab IV at Week 6 with mandatory transition by Week 14.
  Interventions: Drug: Vedolizumab IV; Drug: Vedolizumab SC

INTERVENTIONS:
Drug: Vedolizumab IV — Vedolizumab IV infusion
  Other Names: Entyvio
Drug: Vedolizumab SC — Vedolizumab SC injection
  Other Names: Entyvio

SUMMARY:
Ulcerative Colitis (UC) and Crohn's Disease (CD) are long-term conditions in the gut that can cause diarrhea, swelling (inflammation), bleeding from the anus, and belly pain. The main aim of this study is to check for how many participants with UC and CD signs and symptoms disappear after 3.5 months (14 weeks) of treatment with Vedolizumab (this is called remission).

Participants will be treated with Vedolizumab for approximately 1 year (50 weeks). During the first 1.5 months (6 weeks), participants will receive Vedolizumab as an infusion in the vein (called intravenously). After this, participants will receive Vedolizumab as an injection under the skin (called subcutaneously) for the rest of the treatment. Participants for whom the treatment does not seem to work well after 3.5 months (14 weeks) will stop treatment with Vedolizumab and can change to another treatment and also there will be additional required visits at 6 months (26 weeks) and at 1 year (52 weeks). All participants will be checked again 4.5 months (18 weeks) after their last treatment with Vedolizumab.

During the study, participants will visit their study clinic several times.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this study, participants must meet all the following criteria:

1. In the investigator's opinion, the participant can understand and comply with protocol requirements.
2. The participant signs and dates an electronic informed consent form (ICF) and any required privacy authorization prior to any study procedures.
3. The participant is 18 to 80 years of age at the time of signing the ICF.
4. The participant's immunization is up to date per vedolizumab US prescribing information (USPI).
5. If participant is a woman of childbearing potential (WOCBP):

   1. Agrees to use at least 1 form of highly effective contraception from signing the ICF until at least 18 weeks after the last dose of vedolizumab.
   2. Agrees to avoid donating ova from signing the ICF throughout the duration of the study and for 18 weeks after the last dose of vedolizumab.
   3. Has a negative urine pregnancy test within 3 days before first dose of vedolizumab.
   4. Agrees to forego breastfeeding from first dose of vedolizumab through 18 weeks after the last dose of vedolizumab.
6. If participant is a fertile man:

   1. Agrees to use contraception from signing the ICF until at least 18 weeks after the last dose of vedolizumab
   2. Agrees to avoid donating sperm throughout the study and for 18 weeks after the last dose.
7. The participant has a diagnosis of moderate to severely active UC or CD defined by the following:

   1. CD: A Crohn's Disease Activity Index (CDAI) score of 220 to 450 and a SES-CD >=6 (>=4 if isolated ileal disease) at screening OR
   2. UC: A complete Mayo score (MS) of 6 to 12 with endoscopy subscore of 2 to 3 at screening
8. UC or CD diagnosis established prior to screening by clinical and endoscopic evidence and corroborated by a histopathology report.
9. Demonstrated an inadequate response to, loss of response to, or intolerance of at least one of the following agents: corticosteroids, immunomodulators, and/or advanced therapy.

Exclusion Criteria

Participants who meet any of the following exclusion criteria will be excluded from participation in this study:

1. Received approved or investigational anti-integrin antibodies (i.e., vedolizumab, natalizumab, efalizumab, etrolizumab, abrilumab [AMG 181]) at any time prior to screening.
2. Failed (primary or secondary nonresponse) on more than 2 prior advanced treatments.
3. Use of corticosteroid enemas/suppositories within 2 weeks prior to screening (for UC and CD).
4. In the investigator's opinion the participant meets any contraindication, warnings and precautions, drug interactions, or special population considerations per the vedolizumab USPI, or has (medical history or known allergy, hypersensitivity, or intolerance to vedolizumab or its excipients) (Food and Drug administration [FDA] 2024).
5. Received any investigational biologic therapy <= 6 months prior to screening.
6. The participant has received an advanced treatment for an approved indication other than CD or UC. Advanced therapy include: TNF inhibitors (e.g. infliximab, adalimumab, certolizumab pegol), and IL 12/23 antagonist (e.g. ustekinumab, mirikizumab, risankizumab); and small molecules include JAK inhibitor (e.g. tofacitinib, upadacitinib) and sphingosine-1-phosphate (S1P) receptor modulator (e.g. etrasimod, ozanimod).
7. The participant has any evidence of an active infection during screening.
8. Ileostomy, colostomy, severe, or symptomatic stenosis of the intestine or short bowel syndrome.
9. A surgical procedure requiring general anesthesia within 3 months prior to screening or is planning to or is at risk of undergoing major surgery during the study period.
10. History of malignancy, except for the following: adequately treated nonmetastatic basal cell skin cancer; squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to screening; and history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to screening. Participants with a remote history of malignancy (example, greater than (>) 10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received; this must be discussed with the sponsor on a case-by-case basis prior to enrollment.
11. History of or symptoms of progressive multifocal leukoencephalopathy (PML) in the investigator's opinion.
12. Has laboratory abnormalities during the screening period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of CD Participants With 2-item Patient-reported Outcome Measure (PRO-2) Remission at Week 14 | At Week 14
  PRO-2 remission is defined as 7-day average of very soft or liquid stool frequency (SF) less than and equal to (<=) 2.8, 7-day average of abdominal pain (AP) score <= 1.0, and neither worse than baseline.
Percentage of UC Participants With PRO-2 Remission at Week 14 | At Week 14
  PRO-2 remission is defined as Mayo rectal bleeding sub-score of 0 and stool frequency sub-score <=1.

SECONDARY OUTCOMES:
Percentage of CD and UC Participants With PRO-2 Remission at Weeks 6 and 52 | At Weeks 6 and 52
  PRO-2 remission for CD participants is defined as 7-day average of very soft or liquid SF <= 2.8, 7-day average of AP score <= 1.0, and neither worse than baseline. PRO-2 remission for UC participants is defined as Mayo rectal bleeding sub-score of 0 and stool frequency sub-score <=1.
Percentage of CD and UC Participants With Clinical Response at Weeks 6, 14, and 52 | At Weeks 6, 14, and 52
  CD clinical response is defined as greater than and equal to (>=) 100 points decrease from baseline in CDAI score. UC clinical response is defined as reduction in complete Mayo score of >=3 points and >=30 percent (%) from baseline with an accompanying decrease in rectal bleeding sub-score of >=1 point(s) or absolute rectal bleeding sub-score of <=1 point or absolute rectal bleeding sub-score of <=1 point, or a reduction in partial Mayo score of >=2 points and >=25% from baseline, if complete Mayo score was not performed at visit.
Percentage of CD Participants With Endoscopic Response at Week 52 | At Week 52
  Endoscopic response is defined as >=50% reduction from baseline (or for participants with isolated ileal disease, SES-CD <= 4 or at least a 2-point reduction from baseline) in Simple Endoscopic Score for Crohn's Disease (SES-CD) score. SES-CD evaluates 4 endoscopic variables (the intestinal surface affected by ulcers, the intestinal surface affected by other inflammatory lesions, the presence of ulcers, and the presence of narrowing).
Percentage of CD Participants Achieving Endoscopic Remission at Week 52 | At Week 52
  Endoscopic remission as per SES-CD is defined as SES-CD score <=4 or <=2 for ileal disease, no subscore >1. SES-CD evaluates 4 endoscopic variables (the intestinal surface affected by ulcers, the intestinal surface affected by other inflammatory lesions, the presence of ulcers, and the presence of narrowing).
Percentage of UC Participants With Improvement of Endoscopic Appearance of the Mucosa at Week 52 | At Week 52
  Improvement of endoscopic appearance of the mucosa is defined as Mayo endoscopic sub-score = 0 (normal or inactive disease) or 1 (mild disease [erythema, decreased vascular pattern, mild friability]).
Percentage of UC Participants With Endoscopic Remission at Week 52 | At Week 52
  Endoscopic remission is defined as a centrally read complete Mayo endoscopy subscore of 0.
Percentage of CD and UC Participants With Clinical Remission at Weeks 6, 14, and 52 | At Weeks 6, 14, and 52
  Clinical Remission for CD is defined as a CDAI <150 point. Clinical remission for UC is defined as complete MS of <=2 points and no participant sub-score greater than (>) 1 point or defined as a partial Mayo score (stool frequency, rectal bleeding, physician's global assessment [PGA]) score of <=2 and no individual sub-score >1.
Percentage of CD and UC Participants With Clinical Remission at Week 52 | At Week 52
  Clinical remission for CD is defined as a CDAI <150 point. Clinical remission for UC is defined as complete MS of <=2 points and no participant sub-score >1 point or defined as a partial Mayo score (stool frequency, rectal bleeding, PGA) score of <=2 and no individual sub-score >1. Percentage of CD and UC participants with clinical remission at Week 52, among those participants who achieved clinical remission at Week 6 and 14 will be reported.
Change From Baseline in C-reactive Protein (CRP) levels of CD and UC Participants at Weeks 6, 14, and 52 | Baseline, Weeks 6, 14, and 52
  Change from baseline in CRP levels of CD and UC participants at Weeks 6, 14, and 52 will be reported.
Change From Baseline in Fecal Calprotectin Concentrations of CD and UC participants at Weeks 6, 14, and 52 | Baseline, Weeks 6, 14, and 52
  Change from baseline in fecal calprotectin concentrations of CD and UC participants at Weeks 6, 14, and 52 will be reported.
Number of CD and UC Participants With Serious Infections | Up to end of study (up to 72 weeks)
  Number of CD and UC participants with serious infections will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (85):
- United States (85):
  - Gastro Health Research- St. Vincents East, Birmingham, Alabama
  - East View Medical Research, Mobile, Alabama
  - Spectrum Research Institute LLC, Gilbert, Arizona
  - GI Alliance- Sun City, Sun City, Arizona
  - UAMS Health Gastroenterology Clinic, Little Rock, Arkansas
  - Gastroenterology and Liver Institute, Escondido, California
  - Inland Empire Gastroenterology, Murrieta, California
  - Digestive Health Institute, Newport Beach, California
  - Knowledge Research Center, Orange, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Associates in Gastroenterology, PC, Colorado Springs, Colorado
  - Rocky Mountain Endocopy Centers LLC, Littleton, Colorado
  - Access Research Institute, Brooksville, Florida
  - Gastro Florida, Clearwater, Florida
  - Doral Medical Research, LLC, Hialeah, Florida
  - Digestive and Liver Center of Florida, P.A., Kissimmee, Florida
  - Gastro Health Research - Miami, Miami, Florida
  - The Clinical Trials Network CTNX LLC, Orange City, Florida
  - Endoscopic Research, Inc., Orlando, Florida
  - Orlando Health-Orlando Regional Medical Center, Orlando, Florida
  - Digestive and Liver Center of Florida, Orlando, Florida
  - Gastro Health Research - Pensacola, Pensacola, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Atlanta Gastroenterology Associates LLC, Atlanta, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Yapp, Rockford M.D. (Private Practice), Downers Grove, Illinois
  - GI Alliance - Glenview, Glenview, Illinois
  - Gastroenterology and Internal Medicine Specialists, SC, Lake Barrington, Illinois
  - Suburban Gastroenterology, Naperville, Illinois
  - GI Partners of Illinois - Southwest Gastroenterology, Oak Lawn, Illinois
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Hutchinson Clinic, Hutchinson, Kansas
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - GI Alliance, Metairie, Louisiana
  - Portland Gastroenterology Center, Portland, Maine
  - Capital Digestive Care, Chevy Chase, Maryland
  - Woodholme Gastroenterology, Glen Burnie, Maryland
  - Gastro Health Research - Framingham, Framingham, Massachusetts
  - Lucida Clinical Trials LLC, New Bedford, Massachusetts
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Huron Gastro, Ypsilanti, Michigan
  - MNGI Digestive Health, P.A., Plymouth, Minnesota
  - Delta Gastroenterology and Endoscopy Center, Southaven, Mississippi
  - GI Associates Research, LLC, Columbia, Missouri
  - Mid America Gastro Intestinal Consultants, Kansas City, Missouri
  - St Charles Clinical Research, Weldon Spring, Missouri
  - Advanced Research Institute, Reno, Nevada
  - Presbyterian Health care services, Albuquerque, New Mexico
  - Westchester Putnam Gastroenterology PC, Carmel, New York
  - IMIDeology, Elmhurst, New York
  - NYU Langone Long Island Clinical Research Associates, Lake Success, New York
  - Lenox Hill Hospital, New York, New York
  - New York Gastroenterology Associates, New York, New York
  - Manhattan Clinical Research, LLC, New York, New York
  - Gastroenterology Group of Rochester, Rochester, New York
  - ProHealth (Seaford) (Optum), Seaford, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - Charlotte Gastroenterology and Hepatology, P.L.L.C, Charlotte, North Carolina
  - Pinehurst Medical Clinic Inc, Pinehurst, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - Gastro Health Research - Cincinnati, Cincinnati, Ohio
  - DSI Research Northridge LLC, Dayton, Ohio
  - Gastro Health Research - Liberty Township, Liberty Township, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - DSI Research LLC, Springboro, Ohio
  - NorthShore Gastroenterology Research, LLC, Westlake, Ohio
  - The Oregon Clinic, P.C., Portland, Oregon
  - University Gastroenterology, Providence, Rhode Island
  - Palmetto Primary Care Physician Division of Gastroenterology, Summerville, South Carolina
  - Tri-Cities Gastroenterology, Kingsport, Tennessee
  - The Clinical Trials Network CTNX LLC, El Paso, Texas
  - Amel Med LLC, Georgetown, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Integrity Advanced Therapeutics, Houston, Texas
  - One of a Kind Clinical Research Center LLC, Kingwood, Texas
  - West Texas Research Institute, Lubbock, Texas
  - Texas Gastro Consultants, Tomball, Texas
  - Digestive Research of Central Texas, LLC, Waco, Texas
  - GI Alliance - Webster, Webster, Texas
  - Advanced Research Institute, Ogden, Utah
  - Gastroenterology Consultants of Southwest Virginia., Roanoke, Virginia
  - TMPG Clinical Research, Williamsburg, Virginia
  - GI Alliance, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/6a28167d326b42b3??page=1&idFilter=Vedolizumab-4063